CLINICAL TRIAL: NCT06248801
Title: A Bioequivalence Study of Vildagliptin and Metformin Tablets 50/1000 mg Relative to GALVUS MET (50mg/1000 mg) Tablets in Healthy Thai Adult Volunteers Under Fed Condition.
Brief Title: Vildagliptin and Metformin Tablets 50/1000 mg Relative to GALVUS MET (50mg/1000 mg) Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bio-innova Co., Ltd (Industry)
Responsible Party: Principal Investigator, Sasitorn Kittivoravitkul, Principal Investigator, Bio-innova Co., Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VME-005-22
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Healthy Subjects
Keywords: Bioequivalence Vildagliptin and Metformin tablets 50/1000 mg
MeSH Terms: interventions — Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1-Vildagliptin and Metformin test product and then reference product (Experimental): Participants will receive treatment 1 in period 1 and treatment 2 in period 2. Where treatment 1= Vildagliptin and Metformin tablets 50/1000 mg test product, treatment 2= Vildagliptin and Metformin tablets 50/1000 mg reference product.
  Interventions: Drug: Vildagliptin and Metformin-Test product
- Sequence 1-Vildagliptin and Metformin reference product and then test product (Experimental): Participants will receive treatment 2 in period 1 and treatment 1 in period 2. Where treatment 1= Vildagliptin and Metformin tablets 50/1000 mg test product, treatment 2= Vildagliptin and Metformin tablets 50/1000 mg reference product.
  Interventions: Drug: Vildagliptin and Metformin-Reference product

INTERVENTIONS:
Drug: Vildagliptin and Metformin-Test product — Vildagliptin and Metformin tablets 50/1000 mg manufactured by Mylan Laboratories Limited, India
  Arms: Sequence 1-Vildagliptin and Metformin test product and then reference product
Drug: Vildagliptin and Metformin-Reference product — Vildagliptin and Metformin tablets 50/1000 mg manufactured by NOVARTIS PHARMA PRODUKTIONS GmbH, Germany.
  Arms: Sequence 1-Vildagliptin and Metformin reference product and then test product

SUMMARY:
The study is to compare the rate and extent of absorption of a generic formulation with that of a reference for mulation when given as equal labeled dose. The study will be randomized, open-label, single dose, two way crossover design with two-period, two-treatment and two-sequence under fasting condition and at least 14 days washout period between the doses.

DETAILED DESCRIPTION:
This protocol describes an open labelled, single-dose, randomized, two-period, two-treatment, two-sequence crossover study to investigate the bioequivalence of two formulations of Vildagliptin and Metformin tablets 50/1000 mg manufactured by Mylan Laboratories Limited, India to GALVUS MET (50mg/1000 mg) tablets manufactured by NOVARTIS PHARMA PRODUKTIONS GmbH, Germany.

Single-dose fed pharmacokinetics will be characterized in 48 healthy, adult volunteers, for a total of 48 healthy adult subjects.

Approximately eight milliliter (1 × 8 mL) blood samples will be collected in K3 EDTA tubes at pre-dose and the following times after dosing: at 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 24.00 and 36.00 hours.

The collected blood samples will be transferred into centrifugation room at controlled temperature (2-8°C) and start centrifuged at 4±2°C within 2 hours after blood sample collection. Up to four (4) aliquots of plasma will be added in four pre-labeled cryovials for approximately 1 mL per each cryovial. Two aliquots for analyze vildagliptin and two aliquotes for analyze metformin. Cryovials containing plasma sample will be transferred to deep freezer in controlled temperature (2-8 °C) and will be stored at -70±10 °C.

For the determination of the pharmacokinetic disposition of the formulations, there will be a total of 48 blood samples involving a total of 385 mL (including 10 mL for screening and 7 mL for post-study safety monitoring) of blood collected for pharmacokinetic analysis from each subject who provid their complete all blood collections in the study. There will be at least 7 days between dosing times for the treatment periods.

The bioequivalence of Vildagliptin and Metformin tablets 50/1000 mg manufactured by Mylan Laboratories Limited, India to GALVUS MET (50mg/1000 mg) tablets manufactured by NOVARTIS PHARMA PRODUKTIONS GmbH, Germany will be assessed by a statistical comparison of various pharmacokinetic parameters derived from the plasma concentration-time curves of Vildagliptin and Metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 55 years, Subject must meet age requirements at the time of signing the initial informed consent and the initial study medication administration.
2. Sex: Males and/or non-pregnant, non-lactating females.

   1. Women of childbearing potential must have a negative urine human chorionic gonadotropin (hCG) pregnancy test performed on screening day and prior to the initial dose of each period of study medication.
   2. Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

      1. postmenopausal with spontaneous amenorrhea for at least one (1) year
      2. bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
      3. total hysterectomy and an absence of bleeding for at least 3 months.
3. Weight: Each subject is required to have a Body Mass Index (BMI) value less than or equal to 30.0 kg/m2 but greater than or equal to 18.5 kg/m2. All weight values are to be reported according to the scale's precision. The subject's height is to be reported in centimeters to the nearest tenth. Each subject's BMI is to be calculated using the reported weight in kilograms and height in centimeters and it is to be reported to the nearest tenth (26.3 kg/m2).
4. Smoking Status: Moderate smokers (up to 10 cigarettes or equivalent per day refer to Appendix VII: Nicotine Equivalence Estimates) are permitted.

   • Documentation of smoking status is to be via the questionnaire in Appendix VI, with results included in the study database (if applicable), and Subject's CRF.
5. Adequate venous access in both arms for the collection of a number of blood samples during the study.
6. Able to understand and sign the written Informed Consent Form.

   a. Utilization of illiterate subjects is permitted when performed according to GCP, as well as regulations/guidances for the region of submission and country of conductance.
7. Willing to follow the protocol requirements and comply with protocol restrictions and allow investigators to draw approximately 7 mL of blood for monitoring subjects' safety after the completion of the study.
8. Willing to follow precautions during driving and operating machines
9. All subjects should be judged by the Principal Investigator or Medical Sub-Investigator as normal and healthy during a pre-study medical evaluation performed within 28 days of the initial dose of study medication which will include:

   1. a normal or non-clinically significant physical examination, including vital signs (blood pressure, pulse rate, respiratory rate and forehead-surface temperature)
   2. within normal limits or non-clinically significant laboratory evaluation results for the following tests (unless otherwise noted in the Exclusion Criteria):

      * Serum Chemistries Alkaline Phosphatase Albumin Creatinine AST Blood sugar (by DTX) Total Protein Total Bilirubin ALT Direct Bilirubin BUN
      * Hematology Platelet Count White Blood Cell Count Hemoglobin Hematocrit Red Blood Cell Count Neutrophils Lymphocytes Monocytes Eosinophils Basophils MCV, MCH, MCHC
      * Additional tests may be performed, if necessary, based on standard lab panels utilized by the clinical site.
   3. Normal or non-clinically significant 12-lead EKG
   4. Negative Hepatitis B antigen test
   5. Negative Hepatitis C antibody test
   6. Negative HIV test
   7. Negative urine drug screen including at a minimum Metamphetamines, benzodiazepines, cocaine, opioids and Marijuana (THC),
   8. if tobacco/nicotine use is suspected, a urine cotinine test may be performed at the discretion of the Principal Investigator or responsible physician and if performed, must be negative,
   9. if warranted, other tests and/or examinations may be performed at the discretion of the Principal Investigator or responsible physician.

Exclusion Criteria:

1. Institutionalized subjects.
2. Social Habits:

   1. Consumption of any alcoholic beverage within the 48 hours prior to the initial administration of study medication and until the completion of each period of the study.
   2. Consumption of any caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial administration of study medication and until the completion of each period of the study.
   3. Consumption of seville oranges grapefruit, grapefruit-like, or grapefruit containing products within 48 hours prior to the initial administration of the study medication and until the completion of each period of the study.
   4. Any recent, significant change in dietary or abnormal diet within 48.0 hours prior to dosing.
   5. History of drug and/or alcohol abuse within one year of start of study.
   6. Use of any nicotine containing product within the 7 days of the initial administration of study medication until the completion of the study.
3. Medications

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial administration of study medication.
   2. A depot injection or implant of any drug within 3 months prior to initial administration of study medication.
   3. Use of any medication, vitamin, herbal supplement, or vitamin known to induce or inhibit hepatic enzyme activity within 14 days prior to the initial administration of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, genitourinary, musculoskeletal disease or malignancies unless deemed not clinically significant by the Principal Investigator or Medical Sub-Investigator.
   2. History of tuberculosis.
   3. History of difficulties in swallowing, or any gastrointestinal disease (i.e. cholecystectomy) or previous GI surgery other than appendectomy which could affect drug absorption. History of gastrointestinal obstruction, particularly paralytic ileus.
   4. Acute illness at the time of either the pre-study medical evaluation or dosing period I.
5. Any reason which, in the opinion of the Principal Investigator or Medical Sub-Investigator, would prevent the subject from safely participating in the study.
6. Intolerance to venipuncture.
7. Donation or loss of blood or plasma within 90 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to Vildagliptin, Metformin, other related products, or any inactive ingredients.
9. Subjects who have received an investigational drug within 90 days prior to the initial dose of study medication.
10. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator or Medical Sub-Investigator, could contraindicate the subject's participation in this study.
11. Subject with B.P. is Systolic B.P < 90, ≥140 mm/Hg, Diastolic B.P < 60, ≥90 mm/Hg or pulse rate > 100 beats per minute.
12. Serum bilirubin greater than 1.5 times the upper limit of reference range (ULRR).*
13. Serum creatinine greater than 1.5 times the upper limit of reference range (ULRR).*
14. Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 2 times the upper limit of reference range (ULRR).*
15. Participation in any clinical study within the past 3 months before the study. (* Depend on decision of principal investigator, medical sub-investigator and/or clinical investiagtor)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC 0-t) | Blood samples will be collected for PK analyses in each period pre-dose (0.00 hour) and at 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 24.00 and 36.00 hours post-dose.
  pre-dose (0.00 hour) and at 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 24.00 and 36.00 hours post-dose.
Maximal measured plasma concentration (Cmax) | Blood samples will be collected for PK analyses in each period pre-dose (0.00 hour) and at 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 24.00 and 36.00 hours post-dose.
  pre-dose (0.00 hour) and at 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 24.00 and 36.00 hours post-dose.

SECONDARY OUTCOMES:
Number of subjects with adverse events | Approximately the day 14 after the last visit
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

IPD SHARING:
Plan to Share IPD: No
Company Policy